CLINICAL TRIAL: NCT03936374
Title: A Study to Evaluate the Effect of Coadministration of a Proton Pump Inhibitor (Omeprazole) on the Pharmacokinetics of BMS-986205 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Omeprazole on the Pharmacokinetics of BMS-986205 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CA017-089
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — linrodostat; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986205 + Omeprazole (Experimental)
  Interventions: Drug: BMS-986205; Drug: omeprazole

INTERVENTIONS:
Drug: BMS-986205 — Participants will receive BMS-986205 on Days 1 and 15
Drug: omeprazole — Participants will receive omeprazole on Days 10 to 15

SUMMARY:
The purpose of this study is to assess the effect of multiple dose administrations of Omeprazole on the pharmacokinetics of BMS-986205.

ELIGIBILITY:
Inclusion Criteria:

* Health male and female participants (not of childbearing potential) as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) greater than or equal to (>=) 80 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2)
* Body mass index (BMI) of 18.0 kilogram per meter square (kg/m^2) to 32.0 kg/m^2
* Women participants must have documented proof that they are not of childbearing potential

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding
* Active tuberculosis (TB) requiring treatment or documented latent TB within the previous 3 years
* Concomitant use of strong inhibitors or strong inducers of CYP3A4
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of BMS-986205 | Up to Day 29
Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration [AUC(0-T)] of BMS-986205 | Up to Day 29
Area Under the Plasma Concentration-time Curve from Time Zero Extrapolated to Infinite Time [AUC(INF)] | Up to Day 29

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Discontinuation | Up to Day 36
Number of Participants with Vital Sign Abnormalities | Up to Day 29
Number of Participants with 12-lead Electrocardiogram (ECG) Abnormalities | Up to Day 29
Number of Participants with Physical Examination Abnormalities | Up to Day 29
Number of Participants with Clinical Laboratory Results Abnormalities | Up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Davidson, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls